CLINICAL TRIAL: NCT00263809
Title: Evaluation of the Safety and Performance of Platelet Transfusion Products Treated With MIRASOL® Pathogen Reduction Technology. A Study in Human Thrombocytopenic Subjects.
Brief Title: Safety and Performance of MIRASOL® PRT Treated Platelet Transfusion Products
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Terumo BCTbio (Industry)
Responsible Party: Tracy Roberts, Director of Clinical Affairs, Navigant Biotechnologies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTS-0028
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

ARMS (2):
- 1 (Experimental): Treatment, Mirasol-treated platelets
  Interventions: Device: Pathogen Reduction Technology
- 2 (No Intervention): Reference, Untreated platelets

INTERVENTIONS:
Device: Pathogen Reduction Technology
  Arms: 1

SUMMARY:
The primary objective of the study is to measure platelet corrected count increments and the incidence of serious adverse events (SAE). The primary endpoint is the platelet corrected count increment measured 1-hour post transfusion in response to the infusion of platelet concentrates treated with the Mirasol PRT System device (test product) versus untreated (reference product).

DETAILED DESCRIPTION:
The objective of the study is to determine if the MIRASOL Pathogen Reduction Technology (PRT) System for Platelets device performs safely and maintains adequate platelet performance in a clinical setting. This will be achieved by comparing the platelet corrected count increment measured 1 hour post transfusion and the incidence of serious adverse events in response to the infusion of platelet concentrates treated with the device (test product) versus untreated (reference product) in thrombocytopenic subjects requiring platelet transfusions. The performance, safety, and tolerability profile of the device will be further assessed by monitoring and comparing the incidence of discontinuations due to adverse events in relation to platelet transfusion up to 4 weeks after transfusion, including the incidence of transfusion associated infections, and the number and time between transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age of 16 years or older
* Women of Child Bearing Potential not pregnant
* Subject must have signed and dated the Informed Consent form
* Hospitalized, thrombocytopenic subjects and expected to receive at least two platelets transfusion

Exclusion Criteria:

* History of any hypersensitivity reaction to riboflavin or metabolites
* History of refractoriness to platelet transfusions
* Positive lymphocytotoxic antibody test
* Active bleeding
* Splenomegaly
* Acute or chronic Disseminated Intravascular Coagulation
* History or diagnosis of Immune/Idiopathic Thrombocytopenic Purpura, Thrombotic Thrombocytopenia Purpura, or Haemolytic Uremic Syndrome
* History or diagnosis of an autoimmune disease affecting haemostasis
* History of solid organ transplants
* Evidence of occlusive venous disease
* Clinical signs of infection at the time of inclusion
* Pregnant or lactating females
* Chronic alcohol misuse
* Use of prohibited medications

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The platelet corrected count increment measured 1 hour post transfusion.

SECONDARY OUTCOMES:
The platelet corrected count increment measured 24 hours post-transfusion.
The number of days between platelet transfusions during the period of the study.
The number of platelet transfusions per subject.
The number of platelets infused per subject.
The number of platelets used.
The frequency of refractoriness to platelet transfusion.
In case of refractoriness, the evidence for neoantigen immunization against test product.
The number of red blood cell transfusions during the study period.
The incidence of serious adverse events in relation to platelet transfusions.
The incidence of any adverse events in relation to platelet transfusions.
The occurrence of bleeding episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Cazenave, MD, Principal Investigator — Director - EFS Alsace - France
Locations (10):
- France (10):
  - Centre Hospitalier Universitaire Jean Minjoz, Besançon
  - EFS Bourgogne - Franche-Comté, Besançon
  - EFS Aquitaine, Bordeaux
  - Centre Hospitalier Univesrsitaire A Michallon, La Tronche
  - EFS Rhône-Alpes (Site de Grenoble), La Tronche
  - EFS Pays de la Loire, Nantes
  - Centre Hospitalier Universitaire Hôtel Dieu, Nantes
  - Centre Hospitalier Universitaire de Bordeaux, Pessac
  - Centre Hospitalier Régional Universitaire Hautepierre, Strasbourg
  - EFS Alsace, Strasbourg